CLINICAL TRIAL: NCT00531830
Title: Assessment of Factors Which Predict Improvement in Children With PDD After a Year of Integrative Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Other Study IDs: Children with PDD -31CTIL
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Pervasive Developmental Disorder
Keywords: children with PDD
MeSH Terms: conditions — Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Preschool children with PDD
- 2: Preschool children without PDD

SUMMARY:
The aim of the current research is to assess the efficiency of the Integrative Therapy among children with PDD after a year of treatment in kindergartens in Ashdod, Israel.

An additional aim is to pinpoint specific changes in communication quality and functioning in different areas and recognize the prognostic factors, such as social interaction, affect and level of play. This analysis will contribute to developing more efficient treatment program, adapted to the needs of the treated children.

DETAILED DESCRIPTION:
Integrative Therapy among children with PDD after a year of treatment in kindergartens in Ashdod, Israel.

An additional aim is to pinpoint specific changes in communication quality and functioning in different areas and recognize the prognostic factors, such as social interaction, affect and level of play. This analysis will contribute to developing more efficient treatment program, adapted to the needs of the treated children.

ELIGIBILITY:
Inclusion Criteria:

* Children with PDD
* Children aged from 2 years to 6 years

Exclusion Criteria:

* Children with severe retardation

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Irit Orian, M.D., Principal Investigator — Mental health unit for preschoolers, Ashdod, Israel; Beatriz Priel, Prof., Study Director — Ben Gurion University, Beer-Sheva; Alexander Rejba, M.A., Study Chair — Ben-Gurion University, Beer-Sheva